CLINICAL TRIAL: NCT02780752
Title: Dose Ranging Studies of Oral Hymecromone on Hyaluronan Synthesis
Brief Title: A Study of Oral Hymecromone and Hyaluronan Synthesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paul Bollyky (Other)
Responsible Party: Sponsor-Investigator, Paul Bollyky, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-43805
Record Dates: First submitted 2016-05-17; First posted 2016-05-23 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Healthy; Respiratory Disease
MeSH Terms: conditions — Respiration Disorders | interventions — Hymecromone

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three treatment groups, each including up to 6 participants, with treatment over 4 days of different doses of oral hymecromone. Following a wash-out period, participants are allowed to re-enroll into different treatment groups to provide intra-patient dose comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral hymecromone 400mg po three times per day (Active Comparator): Participants will be administered oral hymecromone 400mg po three times per day (1200 mg)
  Interventions: Drug: hymecromone
- Oral hymecromone 800 mg po three times per day (2400 mg) (Active Comparator): Participants will be be administered oral hymecromone 800 mg po three times per day (2400 mg)
  Interventions: Drug: hymecromone
- Oral hymecromone 1200 mg three times per day (3600 mg) (Active Comparator): Participants will be administered oral hymecromone 1200 mg three times per day (3600 mg)
  Interventions: Drug: hymecromone

INTERVENTIONS:
Drug: hymecromone — Oral Hymecromone
  Other Names: 4-Methylumbelliferone

SUMMARY:
The purpose of this study is to add further understanding to the doses of hymecromone that effectively and safely lead to the inhibition of hyaluronan synthesis. In this study we will investigate both circulating hyaluronan in the serum, as well as tissue hyaluronan, using sputum samples as a non-invasive surrogate.

This is a parallel, open-label, single-center, dose-response study of hymecromone in healthy adults 18 years of age or older. Up to 18 participants will be enrolled. Participants will be treated for 4 days with study drug. Safety as well as biomarkers of pharmacokinetic and pharmacodynamic response will be monitored during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age
* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam
* BMI between 18.5 - 30 kg/m2
* Taking no medications for at least 1 week before and during study enrollment, including drugs of abuse, prescription or OTC medications
* Male subjects who are heterosexually active must use an acceptable method of contraception (abstinence, condom with or without spermicidal agent, or partner contraceptive use as described in requirements for female subjects) to avoid pregnancy in their partner for the entire study period
* Female subjects who are heterosexually active must use an acceptable method of contraception: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, IUD, or Hormone-based contraceptive
* Be able to provide written informed consent and comply with requirements of the study
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 3pm the night before a study day until completion of that study day
* Be able to read, speak and understand English
* Able and willing to understand the study, adhere to all study procedures, and provide written informed consent

Exclusion Criteria:

* Subjects with a history of gastrointestinal disease including gastroesophageal reflux disease, gastritis, peptic ulcer disease or dyspepsia
* Subjects with history of dysphagia, achalasia, or difficulty swallowing capsules, tablets or pills
* Subjects with liver failure or LFTs above the upper limit of normal
* Subjects with clinically significant elevations in SCr, BUN or other screening laboratory tests as determined by study physician
* Subjects with a baseline corrected Fridericia's QT interval (QTcF) >450ms and a baseline ECG abnormalities which in the opinion of the study physician, is clinically significant
* Subjects with ongoing alcohol or illegal drug use
* Subjects who are pregnant, lactating or attempting to conceive
* Known allergy to hymecromone or any component thereof
* Physician concern that participant may not adhere to the study protocol
* Current participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Change in sputum hyaluronan concentration over the study period | From baseline to day 4
Change in serum hyaluronan concentration over the study period | From baseline to day 4
Change in serum hymecromone concentration over the study period | From baseline to day 4

SECONDARY OUTCOMES:
The safety and tolerability (as codified by Common Terminology Criteria for Adverse Events (CTCAE) v5.0) of oral hymecromone over the study period | Through study completion, an average of 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bollyky, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Salman L, Martinez L, Faddoul G, Manning C, Ali K, Salman M, Vazquez-Padron R. Hyaluronan Inhibition as a Therapeutic Target for Diabetic Kidney Disease: What Is Next? Kidney360. 2023 Jun 1;4(6):e851-e860. doi: 10.34067/KID.0000000000000126. Epub 2023 Apr 14. PMID 37055910
- [Derived] Rosser JI, Nagy N, Goel R, Kaber G, Demirdjian S, Saxena J, Bollyky JB, Frymoyer AR, Pacheco-Navarro AE, Burgener EB, Rajadas J, Wang Z, Arbach O, Dunn CE, Kalinowski A, Milla CE, Bollyky PL. Oral hymecromone decreases hyaluronan in human study participants. J Clin Invest. 2022 May 2;132(9):e157983. doi: 10.1172/JCI157983. PMID 35499083